CLINICAL TRIAL: NCT05734612
Title: The Role of Colchicine in Reducing The Rate of Myocardial Reperfusion Injury in Patients With ST-Elevation Myocardial Infarction After Primary Percutaneous Coronary Intervention: Study on NLRP3, ASC, Caspase, and Troponin
Brief Title: The Role of Colchicine in Reducing The Rate of Myocardial Reperfusion Injury
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Birry Karim, SpPD-KKV, dr. Birry Karim, SpPD-KKV, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-09-1046
Record Dates: First submitted 2023-01-11; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Reperfusion Injury, Myocardial
Keywords: Myocardial reperfusion injury; Colchicine
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — Colchicine; Lactose

STUDY DESIGN:
Intervention Model Description: Participants will be grouped into two groups which are intervention group and control group. Patients in the intervention group receive loading dose of colchicine 1 x 2 mg followed by colchicine 2 x 0,5 mg daily for two consecutive days. Patients in the control group receive loading dose of placebo (lactose) 1 x 2 mg followed by lactose 2 x 0,5 mg daily for two consecutive days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Colchicine and placebo (lactose) will be packed in capsules with the same appearance by the pharmacist. The pharmacist will code the capsules containing colchicine or the capsules containing placebo into group A or group B without informing the participant, care provider, investigator, and outcome assessor regarding the content of each group of capsules. Participant, care provider, investigator, and outcome assessor do not know the content of the capsules given to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine (Experimental): Patients in the intervention group receive loading dose of colchicine 1 x 2 mg followed by colchicine 2 x 0,5 mg daily for two consecutive days.
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Patients in the control group receive loading dose of placebo (lactose) 1 x 2 mg followed by lactose 2 x 0,5 mg daily for two consecutive days.
  Interventions: Drug: Placebo (lactose)

INTERVENTIONS:
Drug: Colchicine — Patients in the intervention group receive loading dose of colchicine 1 x 2 mg followed by colchicine 2 x 0,5 mg daily for two consecutive days.
  Arms: Colchicine
Drug: Placebo (lactose) — Patients in the control group receive loading dose of placebo (lactose) 1 x 2 mg followed by lactose 2 x 0,5 mg daily for two consecutive days.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the role of colchicine in reducing the rate of myocardial reperfusion injury in patients with ST-elevation myocardial infarction after primary percutaneous coronary intervention. The main questions it aims to answer are:

* Does colchicine reduce the rate of myocardial reperfusion injury ?
* Does colchicine reduce the concentration of markers of myocardial reperfusion injury (NLRP3, ASC, caspase, and troponin) ?

Participants will

* Be grouped into intervention group and control group blindly. Patients in the intervention group receive loading dose of colchicine 1 x 2 mg followed by colchicine 2 x 0,5 mg daily for two consecutive days. Patients in the control group receive loading dose of placebo (lactose) 1 x 2 mg followed by lactose 2 x 0,5 mg daily for two consecutive days.
* Undergo peripheral blood vein examination before primary percutaneous coronary intervention, after primary percutaneous coronary intervention, 24 hour after primary percutaneous coronary intervention, and 48 hour after primary percutaneous coronary intervention.

Researchers will compare intervention group and control group to see if colchicine reduces the rate of myocardial reperfusion injury and reduces the concentration of markers of myocardial reperfusion injury (NLRP3, ASC, caspase, and troponin) in patients with ST-elevation myocardial infarction after primary percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ST-elevation myocardial infarction based on clinical symptoms, signs, and electrocardiography who undergo primary percutaneous coronary intervention
* Patients aged 18 - 80 years old

Exclusion Criteria:

* Patients with malignancy
* Patients with allergic reaction to colchicine
* Stroke within the last 3 months
* Severe infection (sepsis)
* Chronic kidney disease with eGFR of <30mL/min/1.73m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-04 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
The Rate of Myocardial Reperfusion Injury | Up to 3 days after primary percutaneous coronary intervention
  The rate of hypotension, acute heart failure, arrhythmias, persistent chest pain, or microvascular obstruction up to 3 days after primary percutaneous coronary intervention after primary percutaneous coronary intervention

SECONDARY OUTCOMES:
Activation of NLRP3 in peripheral blood vein measured in counts | 30 minutes before, 30 minutes after, 24 hours after, and 48 hours after primary percutaneous coronary intervention
  Activation of NLRP3 in peripheral blood vein 30 minutes before, 30 minutes after, 24 hours after, and 48 hours after primary percutaneous coronary intervention measured in counts
Concentration of ASC in peripheral blood vein in ng/ml | 30 minutes before, 30 minutes after, 24 hours after, and 48 hours after primary percutaneous coronary intervention
  Concentration of ASC in peripheral blood vein 30 minutes before, 30 minutes after, 24 hours after, and 48 hours after primary percutaneous coronary intervention in ng/ml
Concentration of caspase in peripheral blood vein in pg/ml | 30 minutes before, 30 minutes after, 24 hours after, and 48 hours after primary percutaneous coronary intervention
  Concentration of caspase in peripheral blood vein 30 minutes before, 30 minutes after, 24 hours after, and 48 hours after primary percutaneous coronary intervention in pg/ml
Concentration of troponin in peripheral blood vein in ng/L | 30 minutes before, 30 minutes after, 24 hours after, and 48 hours after primary percutaneous coronary intervention
  Concentration of troponin in peripheral blood vein 30 minutes before, 30 minutes after, 24 hours after, and 48 hours after primary percutaneous coronary intervention in ng/L

CONTACTS AND LOCATIONS:
Overall Officials: Birry Karim, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deftereos S, Giannopoulos G, Angelidis C, Alexopoulos N, Filippatos G, Papoutsidakis N, Sianos G, Goudevenos J, Alexopoulos D, Pyrgakis V, Cleman MW, Manolis AS, Tousoulis D, Lekakis J. Anti-Inflammatory Treatment With Colchicine in Acute Myocardial Infarction: A Pilot Study. Circulation. 2015 Oct 13;132(15):1395-403. doi: 10.1161/CIRCULATIONAHA.115.017611. Epub 2015 Aug 11. PMID 26265659
- [Background] Akodad M, Lattuca B, Nagot N, Georgescu V, Buisson M, Cristol JP, Leclercq F, Macia JC, Gervasoni R, Cung TT, Cade S, Cransac F, Labour J, Dupuy AM, Roubille F. COLIN trial: Value of colchicine in the treatment of patients with acute myocardial infarction and inflammatory response. Arch Cardiovasc Dis. 2017 Jun-Jul;110(6-7):395-402. doi: 10.1016/j.acvd.2016.10.004. Epub 2017 Jan 3. PMID 28065445
- [Background] Mewton N, Roubille F, Bresson D, Prieur C, Bouleti C, Bochaton T, Ivanes F, Dubreuil O, Biere L, Hayek A, Derimay F, Akodad M, Alos B, Haider L, El Jonhy N, Daw R, De Bourguignon C, Dhelens C, Finet G, Bonnefoy-Cudraz E, Bidaux G, Boutitie F, Maucort-Boulch D, Croisille P, Rioufol G, Prunier F, Angoulvant D. Effect of Colchicine on Myocardial Injury in Acute Myocardial Infarction. Circulation. 2021 Sep 14;144(11):859-869. doi: 10.1161/CIRCULATIONAHA.121.056177. Epub 2021 Aug 23. PMID 34420373
- [Background] Vaidya K, Martinez G, Patel S. The Role of Colchicine in Acute Coronary Syndromes. Clin Ther. 2019 Jan;41(1):11-20. doi: 10.1016/j.clinthera.2018.07.023. Epub 2018 Sep 2. PMID 30185392
- [Background] Raju NC, Yi Q, Nidorf M, Fagel ND, Hiralal R, Eikelboom JW. Effect of colchicine compared with placebo on high sensitivity C-reactive protein in patients with acute coronary syndrome or acute stroke: a pilot randomized controlled trial. J Thromb Thrombolysis. 2012 Jan;33(1):88-94. doi: 10.1007/s11239-011-0637-y. PMID 21918905
- [Background] Robertson S, Martinez GJ, Payet CA, Barraclough JY, Celermajer DS, Bursill C, Patel S. Colchicine therapy in acute coronary syndrome patients acts on caspase-1 to suppress NLRP3 inflammasome monocyte activation. Clin Sci (Lond). 2016 Jul 1;130(14):1237-46. doi: 10.1042/CS20160090. Epub 2016 Apr 21. PMID 27129183
- [Background] Vaidya K, Arnott C, Martinez GJ, Ng B, McCormack S, Sullivan DR, Celermajer DS, Patel S. Colchicine Therapy and Plaque Stabilization in Patients With Acute Coronary Syndrome: A CT Coronary Angiography Study. JACC Cardiovasc Imaging. 2018 Feb;11(2 Pt 2):305-316. doi: 10.1016/j.jcmg.2017.08.013. Epub 2017 Oct 18. PMID 29055633
- [Result] Martinez GJ, Robertson S, Barraclough J, Xia Q, Mallat Z, Bursill C, Celermajer DS, Patel S. Colchicine Acutely Suppresses Local Cardiac Production of Inflammatory Cytokines in Patients With an Acute Coronary Syndrome. J Am Heart Assoc. 2015 Aug 24;4(8):e002128. doi: 10.1161/JAHA.115.002128. PMID 26304941